CLINICAL TRIAL: NCT07212322
Title: A Study to Evaluate the Safety and Efficacy of CD19 UCAR-T Cells in Subjects With Autoimmune Diseases
Brief Title: A Study of CD19 UCAR-T Cells in Subjects With Autoimmune Diseases
Acronym: ET-902-AID01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025102
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus; Idiopahic Inflammatory Myopathies; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Sjögren's Syndrome; Antiphospholipid Syndrome; Immune Thrombocytopenia; Systemic Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Sjogren's Syndrome; Antiphospholipid Syndrome; Purpura, Thrombocytopenic, Idiopathic; Scleroderma, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: CD19 UCAR-T cells

INTERVENTIONS:
Drug: CD19 UCAR-T cells — CD19 UCAR-T cells treatment

SUMMARY:
The purpose of this study is to assess the safety and efficacy of CD19 UCAR-T cell therapy in Subjects with autoimmune diseases.

DETAILED DESCRIPTION:
This is a single-center, one-arm, open-label study aiming to evaluate the safety and efficacy of CD19 UCAR-T Cellsin subjects with autoimmune diseases.

The study process is divided into five periods, including screening, lymphodepletion, treatment, DLT observation and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 65 years old;
* Adequate organ functions, defined as follows:

Hematological function [no transfusion and no use of granulocyte colony-stimulating factor (G-CSF) administration within 2 weeks prior to testing]: white blood cells (WBC) ≥3.0×10^9/L, absolute neutrophil count (ANC)≥1.0×10^9/L, platelet count (PLT)≥50×10^9/L (ITP subjects are without restrictions), hemoglobin ≥80 g/L.

Coagulation function: international normalized ratio (INR) ≤ 1.5×upper limit of normal value （ULN）, and activated partial thromboplastin time (APTT) ≤ 1.5×ULN.

Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤3×(ULN), and total bilirubin ≤1.5×ULN. 4)Renal function: serum creatinine ≤1.5×ULN or creatinine clearance (calculated by Cockcroft Gault formula) ≥ 40 ml/min.

Cardiac function: New York Heart Association (NYHA) Grade I or II, and left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography (ECHO), with no pericardial effusion, and no clinically significant abnormalities on12-lead electrocardiogram (ECG).

Pulmonary function: oxygen saturation ≥92% on room air (without supplemental oxygen), no clinically significant pleural effusion.

* Subjects with fertile partners must agree to use effective contraception throughout the treatment period and for 24 months after treatment, and must refrain from donating eggs/sperm for assisted reproduction during this period; Female subjects of childbearing potential (excluding those who have undergone sterilization or ≥12 months of menopause) must have negative urine or blood pregnancy test results during screening.
* Voluntary participates this trial and can comprehend and sign ICF.
* For subjects with moderate to severe refractory Systemic Lupus Erythematosus:

Diagnosed with SLE according to the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for SLE.

Positive for antinuclear antibody (ANA) (titer ≥1:80) and/or anti-dsDNA antibody and/or anti-Sm antibody at screening.

SLEDAI-2000 score ≥8 at screening; if points are attributed for low complement and/or anti-dsDNA antibody, the SLEDAI-2000 clinical symptom score (excluding points for low complement and/or anti-dsDNA antibody) must be ≥6.

A history of at least 6 months of stable standard treatment regimen prior to screening, with failure to achieve LLDAS criteria for at least 2 months before screening. Standard treatment regimen refers to stable use of any of the following medications (alone or in combination):

glucocorticoids, antimalarials, biologics, and other immunosuppressants or immunomodulators.

• For subjects with relapsed/refractory Systemic Systemic Sclerosis: Diagnosed with systemic sclerosis (SSc) according to the 2013 EULAR/ACR classification criteria for SSc.

Classified as diffuse cutaneous or limited cutaneous subtype with a disease duration ≤7 years (from the first occurrence of Raynaud's phenomenon to screening).

If interstitial lung disease (ILD) is present at screening, forced vital capacity (FVC) must be ≥45% of predicted value, or diffusing capacity for carbon monoxide (DLCO) must be ≥40% of predicted value.

Relapsed/refractory is defined as: failure to respond to prior conventional therapy or disease relapse after remission. Conventional therapy refers to the use of glucocorticoids combined with at least one immunosuppressive/immunomodulatory drug for ≥6 months.

• For subjects with refractory Idiopathic Inflammatory Myopathies: Diagnosed with idiopathic inflammatory myopathy (IIM) with a probability ≥55% according to the 2017 EULAR/ACR classification criteria for IIM, and classified as dermatomyositis (DM), immune-mediated necrotizing myopathy (IMNM), or anti-synthetase syndrome (ASyS) based on age at onset, cutaneous and muscle manifestations, laboratory findings, and muscle biopsy characteristics.

Disease activity/severity meets the following criteria: ①Manual Muscle Testing-8 (MMT-8) score ≤141 (total score 150). ②Meets at least two of the following additional abnormal CSMs: Patient Global Assessment of disease activity [based on Visual Analog Scale (VAS)] score ≥2 (range 0-10); Physician Global Assessment of disease activity VAS score ≥2 (range 0-10); Physician Global Assessment of extra-muscular disease activity VAS score ≥2 (range 0-10); HealthAssessment Questionnaire Disability Index (HAQ-DI) score ≥0.25 (range 0-3); At least one muscle enzyme level >1.5 times the upper limit of normal (ULN).

Previous intolerance or inadequate response to glucocorticoids and at least one immunosuppressant or immunomodulator for the aforementioned autoimmune disease, requiring: Treatment with glucocorticoids and at least one immunosuppressant at known effective doses for at least 3 months.

• For subjects with relapsed/refractory Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis: Clinically diagnosed with granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA) according to the definitions established at the 2012 Chapel Hill Consensus Conference (CHCC).

Meet at least one major item or at least three other items in the Birmingham Vasculitis Activity Score (BVAS) version 3.

Test positive for anti-proteinase 3 (PR3-ANCA) antibody or anti-myeloperoxidase (MPO-ANCA) antibody at screening.

Relapsed/refractory is defined as: Relapsed AAV subjects: Disease relapse (defined as: presence of at least one major item or at least three other items in BVAS assessment, or occurrence of 1-2 new other items in two consecutive assessments) after achieving initial efficacy (BVAS score of 0 and glucocorticoid dose ≤7.5 mg/day prednisone or equivalent) following at least 3 months of treatment with glucocorticoids combined with immunosuppressants, with relapse occurring within 12 weeks prior to screening; Refractory AAV subjects: Failure to achieve efficacy (BVAS score of 0 and glucocorticoid dose ≤7.5 mg/day prednisone or equivalent) after at least 3 months of treatment with glucocorticoids combined with immunosuppressants.

• For subjects with active Sjögren's Syndrome: Diagnosed with Sjögren's syndrome (SS) according to the 2016 EULAR/ACR classification criteria.

Unstimulated whole salivary flow rate ≥0.05 mL/min or stimulated whole salivary flow rate ≥0.01 mL/min at screening.

Active disease defined as: EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score ≥5 points.

• For subjects with refractory Antiphospholipid Syndrome: Diagnosed with antiphospholipid syndrome (APS) according to the 2006 Sydney Revised Classification Criteria for APS or the 2023 ACR/EULAR Classification Criteria for APS; Positive for antiphospholipid antibodies (including lupus anticoagulant, anticardiolipin antibodies, and anti-β2 glycoprotein I antibodies) on at least two occasions >12 weeks apart; Presence of at least one non-criteria clinical manifestation, including thrombocytopenia, hemolytic anemia, aPL nephropathy, valvular heart disease, and neurological manifestations.

• For subjects with chronic/refractory Immune Thrombocytopenia: Diagnosed with immune thrombocytopenia (ITP) according to the Chinese Guideline for Diagnosis and Management of Adult Primary Immune Thrombocytopenia (2020 Edition).

Patients who previously received at least one guideline-recommended standard ITP treatment but exhibited inability to maintain response, relapse, intolerance to standard therapy, or insufficient response.

Chronic/refractory definition: Chronic: Persistent thrombocytopenia for ≥12 months; Refractory: Failure to respond to first-line therapies, thrombopoietin receptor agonists, and rituximab; or failure/relapse after splenectomy; with confirmed ITP diagnosis upon recent reassessment.

Exclusion Criteria:

* Patients with a history or concurrent diagnosis of active malignancies, including tumor-associated polymyositis/dermatomyositis, are excluded. Exceptions include cured or non-recurrent cervical carcinoma in situ for at least 3 years, non-invasive basal cell or squamous cell skin cancer, or localized prostate cancer treated with radical therapy, or ductal carcinoma in situ after radical surgery.
* Patients who have previously received CD19-targeted drugs, or CAR-T therapy, or any other gene therapy products.
* Patients with severe pulmonary diseases within the past year, such as moderate to severe pulmonary hypertension (pulmonary artery systolic pressure > 50 mmHg on echocardiography), or those requiring oxygen therapy via a reservoir mask or non-invasive/invasive mechanical ventilation during screening.
* Patients who have received any of the following medications or treatments within the specified timeframes:

B-cell-depleting therapy within 6 months before screening, assessed by the investigator as not having failed treatment, including anti-CD20, anti-CD22, anti-CD52, anti-CD38 or ant-BCMA monoclonal antibodies or bispecific antibodies.

High-dose intravenous immunoglobulin (IVIG) within 3 months before screening. Dialysis or plasmapheresis within 2 months before screening. Glucocorticoid pulse therapy (defined as ≥ 200 mg/day prednisone or equivalent doses of other glucocorticoids) within 2 months before screening.

Used telitacicept within 6 weeks before screening, or belimumab within 8 weeks before screening.

Thrombopoietin (TPO) or TPO receptor agonists (TPO-RA) or any other medication with a clearly indicated platelet-boosting effect, ortransfusion therapy (including platelet transfusion) within 2 weeks before screening (ITP subjects are without restrictions).

* Patients with a history of severe central nervous system (CNS) disorders history or related symptoms (excluding isolated trigeminal nerve disease) within the past 6 months, including but not limited to: lupus encephalopathy, cerebrovascular diseases, encephalitis, brain injury, aneurysm, cerebellar disorders, organic brain syndrome, Parkinson's disease as well as symptoms such as epilepsy, convulsion, aphasia, dementia.
* Complicated with severe renal disease, defined as any of the following within 8 weeks before screening:

Severe lupus nephritis [defined as urine protein > 6g/24h or serum creatinine > 1.5×ULN.

Creatinine clearance (Cockcroft Gault formula) < 40mL/min]. Active nephritis requiring treatment that are prohibited per protocol. Requiring hemodialysis or plasmapheresis, or receiving prednisone > 100mg/d or equivalent corticosteroid therapy ≥14 days.

* Patients with severe allergies to any components of the lymphodepletion regimen or CD19 UCAR-T therapy used in this study.
* Patients who meet any of the following criteria:

Positive for hepatitis B surface antigen (HBsAg) AND positive for hepatitis B core antibody (HBcAb) with detectable HBV DNA in peripheral blood.

Positive for hepatitis C virus (HCV) antibody with detectable HCV RNA. Positive for Treponema pallidum antibody. Positive for HIV antibody.

* Patients with uncontrolled fungal, bacterial, or viral infections, or any other active infections are assessed as inappropriate to participate in the study by investigator .
* Patients with a history of major organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
* Patients with active tuberculosis (TB) or latent TB infection (defined as positive tuberculin skin test or interferon-gamma release assay results without clinical symptoms or radiographic evidence) at screening;
* Patients who have experienced any of the following cardiovascular events within 6 months before screening (including but not limited to):

Congestive heart failure, myocardial infarction, unstable angina, coronary angioplasty, stenting, coronary/peripheral artery bypass grafting.

Severe arrhythmias requiring treatment (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsade de pointes, etc.). Congenital long QT syndrome and left anterior fascicular block (bifascicular block). Asymptomatic right bundle branch block is permitted for enrollment.

Uncontrolled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure >100 mmHg), history of hypertensive crisis or hypertensive encephalopathy;

* Patients with a history of autoimmune diseases (other than the target indications) that need systemic treatments, including but not limited to: eosinophilic granulomatous with polyangiitis (EGPA), Henoch-Schönlein purpura (HSP), rheumatoid arthritis, cryoglobulinemia vasculitis, inclusion body myositis, anti-glomerular basement membrane disease, Behcet's disease or Takayasu's arteritis, etc..
* Patients with non-IIM conditions such as drug-induced myopathy, HIV-associated myopathy, thyroid myopathy, or a family history of myopathy.
* History of catastrophic APS within 3 months prior to screening;
* Pregnant or lactating women.
* Patients who have received live vaccines within 6 weeks prior to lymphodepleting chemotherapy.
* Patients who meet any of the following criteria:

Participate in other interventional clinical studies, and receipt of any investigational treatment within 3 months before signing the informed consent form.

Intent to participate in another clinical trial during the entire study period. Plan to receive non-protocol-specified treatments for autoimmune diseases.

* Patients with psychiatric disorders including depression or suicidal tendency.
* Patients deemed by the investigator to have other factors that may make them unsuitable for participation or may affect their ability to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Time Frame: 0~28 day after treatment
Frequency of AEs, SAEs | Time Frame: from lymphodepletion to 12 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No